CLINICAL TRIAL: NCT02311647
Title: Uterine Cavity Assessment and Endometrial Gene Expression in Tamoxifen Treated Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-1374-SD-CTIL
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Endometrial Receptivity Post Tamoxifen Exposure
Keywords: Tamoxifen; Uterine cavity; endometrium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post Tamoxifen exposure group: Breast cancer patients receiving or formerly received Tamoxifen for at least 1 year.
- Control group: Breast cancer patients who did not receive endocrine treatment

SUMMARY:
The aim of this multi-center study is to assess the effects of Tamoxifen on the uterine cavity and endometrial abnormalities in young premenopausal women diagnosed with breast cancer.

The research contains two parts: a clinical study and a laboratory study.

* Clinical part: to evaluate the association between tamoxifen treatment and uterine abnormalities.
* Laboratory part: to investigate the effect of Tamoxifen treatment on endometrial tissue, by exploring the molecular aspect of endometrial receptivity.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent malignancy amongst women and approximately 13% of newly diagnosed breast cancer patients are diagnosed between the ages 20-34 [1]. At this age group women are at the peak of their reproductive years, and many have not yet completed family planning. Moreover the age at first birth has steadily increasing in developed nations [2] and more than a quarter of the deliveries are in women above the age of 35. Despite repeated reports in the literature of a worse prognosis in young breast cancer patients, newer treatments have none-the-less improved the outcome amongst young women and for some early stage disease subtypes the outcome is similar to that of older women [3,4]. These increasing numbers of breast cancer survivors are concerned with post-cancer quality of life issues, such as the ability to have children after completing treatment [5-6], hence it is critical to discuss fertility preservation and the ability to conceive when breast cancer is diagnosed [7-9].

Treatment for early breast cancer involves local therapy that includes surgery and adjuvant radiation therapy as well as systemic therapies including chemotherapy, biological therapy and hormonal therapy. Chemotherapy protocols for breast cancer include different combinations of alkylating agents, platinum derivates and taxanes that are toxic to the ovaries, destroy primordial follicle stockpiles, which directly represent ovarian reserve and can result in infertility and premature menopause [10-12].

Tamoxifen Citrate, a Selective Estrogen Receptor Modulator (SERM), competes with estrogen for binding sites in the Estrogen Receptor (ER) in target tissues such as breast. The drug has been in use for over 30 years with a proven high therapeutic index and significant efficacy. The drug is effective in reducing breast cancer recurrence and improving patient's survival across all age groups. The drug is effective in young pre-menopausal breast cancer patients [13-15] . Recently, it has been reported (16) that breast cancer survivors who take tamoxifen for ten years have half the risk of dying from estrogen receptor positive breast cancer. Therefore the new ASCO (American Society of Clinical Oncology ) recommendations are to increase the period of tamoxifen treatment.

However, at this period these patients cannot conceive, in order to enable pregnancy patients should hold Tamoxifen treatment, either with complete termination, or (a more suitable option with the new recommendations) a tamoxifen free window to allow pregnancy should be offered. If ovarian function is preserved women can try to get a spontaneous pregnancy. In patients that suffer from ovarian failure post chemotherapy treatments or embryos (or eggs) that were stored at diagnosis during fertility preservation procedure can be used.

Pregnancies post (and even during) tamoxifen treatment are reported but former breast cancer patients achieve lower pregnancy rate when performing embryo transfer with embryos that were frozen prior to treatment. The chances to conceive post tamoxifen treatments and even more with prolong Tamoxifen treatments are not determined. This becomes of major importance when a limited window of time is allowed for conception.

The risk of developing endometrial cancer for post-menopausal women taking tamoxifen is well established as well as the incidence of endometrial thickening endometrial adhesions and polyps (17). There is no available data whether changes in the endometrium that may be induced by Tamoxifen further impairs the ability to conceive. Ultrasound assessments of the endometrium in patients treated with tamoxifen are limited and often inconclusive mainly due to sub-endometrial ultrasonographic findings that impair evaluation. The incidence of endometrial adhesions and polyps in premenopausal breast cancer patients treated with tamoxifen is unknown. However these abnormalities can interfere with the success of future conception.

The human endometrium is a dynamic tissue that undergoes physiological and clinical changes during the menstrual cycle. Adhesion of the embryo to the endometrium is possible only during a very short period of time, during which the endometrium acquires a functional ability and becomes receptive. This functionality is a pre- requisite for a successful pregnancy.

It is assumed that inadequate uterine receptivity is responsible for approximately two-thirds of implantation failure. Although many fertility disorders have been overcome by a variety of assisted reproductive techniques, implantation remains the rate-limiting step for the success of in vitro fertilization.

As mentioned previously, Tamoxifen may affect the endometrium, however there is no study regarding the effects of these changes on the chances to become pregnant.

Furthermore, tamoxifen effects on endometrial receptivity have not been investigated yet. Although to date no single, clinically relevant morphologic, molecular, or histologic marker capable of indicating endometrial receptivity status has been identified. Few genes were found to be associated with implantation and could act as potential markers for receptivity and can be used to compare endometrial receptivity in patients previously treated with Tamoxifen to normal population. The research will use several genes that have been proven to have high correlation with implantation process and endometrial receptivity.

Aims of the study:

The aim of this multi-center study is to assess the effects of Tamoxifen on the uterine cavity and endometrial abnormalities in young premenopausal women diagnosed with breast cancer.

The research contains two parts: a clinical study and a laboratory study.

* In the clinical part our goal is to evaluate the association between tamoxifen treatment and uterine abnormalities.
* The laboratory study's target is to investigate the effect of Tamoxifen treatment on endometrial tissue, by exploring the molecular aspect of endometrial receptivity

ELIGIBILITY:
Inclusion Criteria:

Breast cancer patients who are:

* < 45 years
* premenopausal
* Had no previous uterine operations (previous D&C is allowed)
* Currently receiving or having received Tamoxifen for at least 1 year.

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Breast cancer patients who are:
  * < 45 years
  * premenopausal
  * Had no previous uterine operations (previous D&C is allowed)
  * Currently receiving or having received Tamoxifen for at least 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Endometrial cells gene expression post Tamoxifen exposure | 2 years

SECONDARY OUTCOMES:
Endometrial thickness post Tamoxifen exposure | 2 Years
Endometrial polyps post Tamoxifen exposure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dror Meirov, MD, Study Director — Sheba Medical Center
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel